CLINICAL TRIAL: NCT01579279
Title: A Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled Study Comparing the Analgesic Efficacy and Safety of ABT-652 to Placebo in Subjects With Diabetic Neuropathic Pain
Brief Title: A Study Comparing the Efficacy and Safety of ABT-652 to Placebo in Subjects With Diabetic Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Stopped
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-210; 2011-003939-56 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-17 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-08

CONDITIONS: Diabetic Neuropathic Pain
Keywords: Diabetic neuropathic pain; Active controlled phase 2 study
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ABT-652 6 mg (Experimental): ABT-652 capsules - twice daily
  Interventions: Drug: ABT-652 6 mg
- ABT-652 12 mg (Experimental): ABT-652 capsules twice daily
  Interventions: Drug: ABT-652 12 mg
- ABT-652 12 mg - 18 mg (Experimental): ABT-652 capsules twice daily
  Interventions: Drug: ABT-652 12 mg - 18 mg
- Placebo (Placebo Comparator): Placebo capsules twice daily
  Interventions: Drug: Placebo
- Duloxetine (Active Comparator): Duloxetine capsules once daily
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: ABT-652 6 mg — 6 mg capsules
  Arms: ABT-652 6 mg
Drug: ABT-652 12 mg — 12 mg capsules
  Arms: ABT-652 12 mg
Drug: ABT-652 12 mg - 18 mg — 12 mg - 18 mg capsules
  Arms: ABT-652 12 mg - 18 mg
Drug: Placebo — Placebo capsules
  Arms: Placebo
Drug: Duloxetine — Duloxetine capsules
  Arms: Duloxetine

SUMMARY:
To evaluate the safety and efficacy of ABT-652 compared to Placebo in subjects with diabetic neuropathic pain. People with diabetes can, over time develop nerve damage throughout the body with symptoms such as pain, tingling, or numbness (loss of feeling) in the hands, arms, feet and legs.

DETAILED DESCRIPTION:
A double blind, randomized, active- and placebo-controlled 13-week study. Duloxetine is added to evaluate assay sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18-75 years with a diagnosis of diabetes mellitus and must have a diagnosis of painful distal symmetric diabetic polyneuropathy and presence of ongoing pain due to diabetic peripheral neuropathy for at least 6 months.
* Subject must have a mean average score of greater than 4 on the 24 hour average pain score (0-10 numerical rating scale) prior to the Baseline Visit.
* Subject has been on a medication for diabetic neuropathic pain for the past 3 months.

Exclusion Criteria:

* Subject has clinically symptomatic neuropathic pain conditions that cannot be distinguished from Diabetic Neuropathic Pain or interfere with the pain assessments of Diabetic Neuropathic Pain.
* A subject has newly diagnosed or clinically significant medical conditions or mental disorders that would preclude participation or would interfere with Diabetic Neuropathic Pain assessments or other functions.
* Subject has clinically significant abnormalities in clinical laboratory tests.
* Subject has taken an opioid chronically, excluding tramadol within the last 3 months prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
24-hour Average Pain Score | 12 weeks
  Weekly mean of 24-hour average pain score measured by a 11-point Numeric Rating Scale completed on subject's daily diary.

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory | 12 weeks
  Measures severity of common neuropathic pain qualities (burning, pressure, squeezing)
Patient Global Impression of Change | 12 weeks
  Captures the subject's evaluation of his/her overall general impression of feeling since beginning study medication
Brief Pain Inventory | 12 weeks
  Capture the subject's severity of pain and interference
Neuropathic Pain Impact on Quality of Life Questionnaire | 12 weeks
  Captures the subject's assessment of neuropathic pain and the effect it has on the quality of daily life
EuroQuality of Life - 5 Dimension -5 Level | 12 weeks
  Capture's the subject's mobility, self-care, usual activity, pain/discomfort and anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Nothaft, MD, Study Director — AbbVie
Locations (8):
- United States (8):
  - Site Reference ID/Investigator# 62887, Anaheim, California
  - Site Reference ID/Investigator# 62824, Walnut Creek, California
  - Site Reference ID/Investigator# 63710, Milford, Connecticut
  - Site Reference ID/Investigator# 62884, DeLand, Florida
  - Site Reference ID/Investigator# 62826, Orlando, Florida
  - Site Reference ID/Investigator# 63703, Brockton, Massachusetts
  - Site Reference ID/Investigator# 73913, Olive Branch, Mississippi
  - Site Reference ID/Investigator# 62886, Dallas, Texas